CLINICAL TRIAL: NCT01413724
Title: Survey of Postoperative Pain and Pain Management in Norwegian Hospitals
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Norwegian Pain Association (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2010/747a
Record Dates: First submitted 2010-07-22; First posted 2011-08-10 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-08

CONDITIONS: Pain, Postoperative
Keywords: Administered analgesic therapy
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Surgical patients: PAtients who had surgery the previous day and are still hospitalized

SUMMARY:
The study is a national survey of pain and pain management to surgical patients in Norwegian Hospitals. Data on pain management are gathered from patient records and data on pain and patient satisfaction are gathered as patients' self report.

ELIGIBILITY:
Inclusion Criteria:

* Surgery previous day

Exclusion Criteria:

* Declined participation
* Unable to communicate (delirious, sedated, intubated)
* Does not read and speak Norwegian
* Patient not available (for instance having physiotherapy og examinations during data collection)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who had surgery the previous day and still are hospitalized. Patients must give informed consent to participate.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2010-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
pain | 24 hours
  Proportion of patients who report average pain intensity >3 on 11 point pain Numerical Rating scale for the first 24 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Olav M Fredheim, MD, PhD, MBA, Principal Investigator — Norwegian University of Science and Technology

REFERENCES:
- [Result] Fredheim OM, Kvarstein G, Undall E, Stubhaug A, Rustoen T, Borchgrevink PC. [Postoperative pain in patients admitted to Norwegian hospitals]. Tidsskr Nor Laegeforen. 2011 Sep 20;131(18):1763-7. doi: 10.4045/tidsskr.10.1129. Norwegian. PMID 21946593
- [Result] Fredheim OM, Borchgrevink PC, Kvarstein G. [Post-operative pain management in hospitals]. Tidsskr Nor Laegeforen. 2011 Sep 20;131(18):1772-6. doi: 10.4045/tidsskr.10.1184. Norwegian. PMID 21946595